CLINICAL TRIAL: NCT06636045
Title: Effect of Blood Flow Restriction (BFR) on Rehabilitation Protocols Following Anterior Cruciate Ligament Reconstruction (ACLR) With Quadricep Autograft
Brief Title: Blood Flow Restriction Following ACLR w/Quad Autograft
Acronym: BFR Quad Delay
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Vopat, Assistant Professor, Orthopedic Surgery, University of Kansas Medical Center
Other Study IDs: UKansasMCRI
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-08

CONDITIONS: Autografts; Blood Flow Restriction Therapy; Rehabilitation Outcome; Quadriceps Muscle Strength; Anterior Cruciate Ligament Reconstruction
Keywords: blood flow restriction; anterior cruciate ligament reconstruction; quadriceps muscle strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BFR Group: Blood Flow Restriction (BFR) will be administered in conjunction with regular physical therapy exercises. BFR training will begin as early as 2 weeks post-op. For 2-3 times/week, as indicated by the patient's physical therapist. This is part of standard practice. Each session will consist of 4 sets (30, 15, 15, and 15 reps) at 80% limb occlusion pressure.
  Interventions: Other: Not applicable- observational study
- Control Group: This group will perform physical therapy without the use of BFR
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — No intervention. Observational study.

SUMMARY:
This project is intended to acquire objective measurements of implementing BFR rehabilitation in ACL reconstructions to show any changes upon completion of the BFR protocol. The results in this study will hopefully represent valuable data in the support of using autografts for ACL reconstructions in high level athletes wanting a full recovery and return to high level of sport.

It has been speculated that use of autografts in ACL reconstructions leads to more quad weakness and muscle atrophy due to tendon harvesting. (Slone et al., 2015) More recently, BFR has shown promise in expediting the recovery and rehabilitation process post-surgically. By implementing BFR following ACL reconstructions with autografts, we hope to mitigate the major deterrent for autograft use and giving patients a more cost-effective approach to surgery. (Hughes et al., 2019)

DETAILED DESCRIPTION:
Specific Aim 1 will identify the overall preservation of muscle and changes in body composition after injury and throughout surgical rehabilitation in athletes undergoing ACL reconstruction. It is hypothesized that implementing BFR rehabilitation protocols following ACL reconstruction with autografts will expedite recovery and return to sport and rescue of muscle tissue at the donor site.

Specific Aim 2 will monitor muscle strength and activation following ACL reconstruction with performance of standardized assessments at intervals. It is hypothesized that BFR implementation will show greater return to strength and enhanced muscle activation during testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing anterior cruciate ligament construction utilizing a quadriceps autograft
* Age 14 - 40 years old

Exclusion Criteria:

* Comorbid conditions (i.e.: hypertension, diabetes, obesity, etc.)
* Patient taking blood thinners or at risk of embolism
* Revision anterior cruciate ligament construction
* Allograft based reconstruction
* Non-quadriceps graft

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject population will be patients of the University of Kansas Health System
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quad muscle Strength | At 6 week post surgical timepoints
  Compare the muscle strength gain or loss between BFR group and control group
Return to sport | 6 week intervals
  Compare the time it takes participants to return to sport in BFR group to control group

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Vopat, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified and compiled prior to analysis, therefore no individual data will be shared.

REFERENCES:
- [Background] Das A, Paton B. Is There a Minimum Effective Dose for Vascular Occlusion During Blood Flow Restriction Training? Front Physiol. 2022 Apr 8;13:838115. doi: 10.3389/fphys.2022.838115. eCollection 2022. PMID 35464074
- [Background] Lu Y, Patel BH, Kym C, Nwachukwu BU, Beletksy A, Forsythe B, Chahla J. Perioperative Blood Flow Restriction Rehabilitation in Patients Undergoing ACL Reconstruction: A Systematic Review. Orthop J Sports Med. 2020 Mar 25;8(3):2325967120906822. doi: 10.1177/2325967120906822. eCollection 2020 Mar. PMID 32232065
- [Background] Hughes L, Rosenblatt B, Haddad F, Gissane C, McCarthy D, Clarke T, Ferris G, Dawes J, Paton B, Patterson SD. Comparing the Effectiveness of Blood Flow Restriction and Traditional Heavy Load Resistance Training in the Post-Surgery Rehabilitation of Anterior Cruciate Ligament Reconstruction Patients: A UK National Health Service Randomised Controlled Trial. Sports Med. 2019 Nov;49(11):1787-1805. doi: 10.1007/s40279-019-01137-2. PMID 31301034
- [Background] Slone HS, Romine SE, Premkumar A, Xerogeanes JW. Quadriceps tendon autograft for anterior cruciate ligament reconstruction: a comprehensive review of current literature and systematic review of clinical results. Arthroscopy. 2015 Mar;31(3):541-54. doi: 10.1016/j.arthro.2014.11.010. Epub 2014 Dec 25. PMID 25543249
- [Background] Sim K, Rahardja R, Zhu M, Young SW. Optimal Graft Choice in Athletic Patients with Anterior Cruciate Ligament Injuries: Review and Clinical Insights. Open Access J Sports Med. 2022 Jul 1;13:55-67. doi: 10.2147/OAJSM.S340702. eCollection 2022. PMID 35800660
- [Background] Cognetti DJ, Sheean AJ, Owens JG. Blood Flow Restriction Therapy and Its Use for Rehabilitation and Return to Sport: Physiology, Application, and Guidelines for Implementation. Arthrosc Sports Med Rehabil. 2022 Jan 28;4(1):e71-e76. doi: 10.1016/j.asmr.2021.09.025. eCollection 2022 Jan. PMID 35141538
- [Background] Castle JP, Tramer JS, Turner EHG, Cotter D, McGee A, Abbas MJ, Gasparro MA, Lynch TS, Moutzouros V. Survey of blood flow restriction therapy for rehabilitation in Sports Medicine patients. J Orthop. 2023 Mar 13;38:47-52. doi: 10.1016/j.jor.2023.03.007. eCollection 2023 Apr. PMID 36969302
- [Background] Tang N, Eren M, Gurpinar T, Ozturkmen Y. A prospective randomized controlled study of hamstring and bone-free quadriceps tendons autografts in arthroscopic ACL reconstruction. Eur J Orthop Surg Traumatol. 2024 Jan;34(1):293-301. doi: 10.1007/s00590-023-03636-5. Epub 2023 Jul 19. PMID 37468645
- [Background] Mistry H, Metcalfe A, Colquitt J, Loveman E, Smith NA, Royle P, Waugh N. Autograft or allograft for reconstruction of anterior cruciate ligament: a health economics perspective. Knee Surg Sports Traumatol Arthrosc. 2019 Jun;27(6):1782-1790. doi: 10.1007/s00167-019-05436-z. Epub 2019 Mar 14. PMID 30874836
- See also: online sample size calculator — https://www.sealedenvelope.com/power/continuous-superiority